CLINICAL TRIAL: NCT02296697
Title: Comparison Between the Effects of Low-level Laser Therapy, High Frequency and Wound Dressing on Pressure Ulcers Treatment: a Clinical Randomized Trial
Brief Title: Low-level Laser Therapy Versus High Frequency on Pressure Ulcers Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 140372
Record Dates: First submitted 2014-10-17; First posted 2014-11-20 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Pressure Ulcer
Keywords: Pressure Ulcer; Low Level Laser Therapy; Dressings
MeSH Terms: conditions — Pressure Ulcer | interventions — Bandages; Saline Solution

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low-level laser therapy AlGaInP (Active Comparator): AlGaInP 660 nm laser and dose of 6 J / cm 2 with point application on the edges of the lesion and sweep up application in the center.
  Interventions: Device: Low-level laser therapy AlGaInP; Other: Wound dressing with saline solution
- High-frequency therapy with O3 formation (Active Comparator): High frequency generator, spherical electrode. Direct spark technique will be used, in which the electrode is positioned millimeters away from the skin of the patient, causing the formation of sparks, with increasing intensity up to 80 to 100% for ozone formation.
  Interventions: Device: High-frequency therapy with O3 formation; Other: Wound dressing with saline solution
- Wound dressing with saline solution (Placebo Comparator): Wound dressing with hygiene of the pressure ulcer with warm saline and after applying the bandage will be held will be held.
  Interventions: Other: Wound dressing with saline solution

INTERVENTIONS:
Device: Low-level laser therapy AlGaInP — Pressure ulcers will be treated with AlGaInP 660 nm laser, wich will be used once a day, five days per week, dosed with 6 J/cm2. Laser therapy is applied punctually in each 1cm2 of the ulcer.
  Other Names: Low-level laser therapy AlGaInP wavelength of 660 nm
  Arms: Low-level laser therapy AlGaInP
Device: High-frequency therapy with O3 formation — High-frequency laser therapy will be applied with spherical electrode, wich contains neon gas inside, from a short distance from the pressure ulcer. The application will last 15 minutes, with increasing intensity from 80 to 100% for ozone formation, once a day, five days per week.
  Other Names: High-frequency therapy with ozone formation
  Arms: High-frequency therapy with O3 formation
Other: Wound dressing with saline solution — Wound dressing will be done daily on patients from the three groups during the study period. On patients who will receive laser therapy and high frequency, the pressure ulcer will be sanitized with worm saline solution in order to clean the wound. This cleaning will be done before and after the interventions.

SUMMARY:
Patients admitted in the Emergency Service that have pressure ulcers will be selected by eligibility criteria and randomized into three groups according to the adopted therapy: wound dressing (CG); wound dressing + high-frequency generator group (GAF); and wound dressing + low-level laser therapy group (GLBP).

DETAILED DESCRIPTION:
Wound dressing is considered the standard treatment for pressure ulcers, however, despite its proven efficacy, it's a long-term healing process. Among Physiotherapy resources available for pressure ulcers treatment, the most used are low-level laser therapy and high-frequency generator. Even though the individual effects of both are evidenced on literature, there are no randomized clinical trials evidencing the effects of low-level laser therapy and high-frequency generator in comparison to wound dressing on pressure ulcers treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pressure ulcers with rate II or III;
* Not receiving pressure ulcer treatment.

Exclusion Criteria:

* Presence of necrotic tissue needing debridement
* Pregnancy
* Discomfort during treatment
* Pressure ulcers with area bigger than 30cm2
* Extensive tunneling
* Diabetes mellitus (DM)
* Severe metabolic disease
* Use of corticosteroids or vasopressors
* Immunosuppression
* Pacemaker
* Neoplasia
* Hemorrhage
* Sensibility disorders
* Metalic device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Changes on pressure ulcer area 28 days after first intervention | Patients will be evaluated on the 7th, 14th, 21st and 28th day after randomized, while hospitalized. If discharge before, follow up will be done untill the last day of hospitalization.
  Evaluated through absolute (mm ²) reduction according to baseline. The participants will be followed while hospitalized, and outcome measure will be assessed at 7th, 14th, 21st and 28th day after the study randomization.

SECONDARY OUTCOMES:
Changes on clinical evolution of the pressure ulcer 28 days after first intervention | Patients will be evaluated on the 7th, 14th, 21st and 28th day after randomized, while hospitalized. If discharge before, follow up will be done untill the last day of hospitalization.
  Clinical evolution of UP through PUSH score. The participants will be followed while hospitalized, and outcome measure will be assessed at 7th, 14th, 21st and 28th day after the study randomization.
Changes on pressure ulcer relative area 28 days after first intervention | Patients will be evaluated on the 7th, 14th, 21st and 28th day after randomized, while hospitalized. If discharge before, follow up will be done untill the last day of hospitalization.
  Evaluated through relative (%) reduction according to baseline. The participants will be followed while hospitalized, and outcome measure will be assessed at 7th, 14th, 21st and 28th day after the study randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Graciele Sbruzzi, Dra, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided